CLINICAL TRIAL: NCT04558762
Title: Ten Years Follow-up, Efficacy and Complications, After Insertion of a MUS Due to Stress Urinary Incontinence, According to the Swedish National Quality Register of Gynecological Surgery.
Brief Title: Ten Years Follow-up After Insertion of a MUS (Mid Urethral Sling) Due to Stress Urinary Incontinence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Stockholm South General Hospital (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Marion Ek, Senior Consultant, Stockholm South General Hospital
Other Study IDs: MUS and SUI
Record Dates: First submitted 2020-09-04; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women who had a MUS inserted.: Women who underwent surgery with insertion of a MUS due to SUI 2006-2010 in Sweden with the MUS coming out retropubic (TVT) or through foramen obturatorium (TOT).
- Controls: Women who have not had a MUS inserted due to stress urinary incontinence. Matched in age.

SUMMARY:
The investigators intend to investigate the long-term complications and the subjective well-being among women who underwent insertion of a MUS due to stress urinary incontinence 2006-2010.

ELIGIBILITY:
Inclusion Criteria:

* Underwent a MUS in Sweden 2006-2010 due to stress urinary incontinence.
* Were registered in The Swedish National Quality Register of Gynecological Surgery.

Exclusion Criteria:

* Did not undergo MUS surgery in Sweden 2006-2010 due to stress urinary incontinence, except those constituting the control group.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who underwent MUS surgery in Sweden 2006-2010 due to stress urinary incontinence.
  The controlgroup will consist of women who did not undergo this surgery but are matched in age with the women who underwent surgery.
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Stress urinary incontinence | +10 years after surgery
  We will measure the percentage of women who suffer from a subjective feeling of stress urinary incontinence ten years after surgery. We will use validated scales; UDI-6 ( Urogenital Distress Inventory), IIQ-7 (Incontinence Impact Questionnaire).

SECONDARY OUTCOMES:
Number of participants with late post operative complications | +10 years after surgery
  Late complications due to surgery such as erosion of the mesh. We will send questionnaires to all participants concerning late post operative complications and we will ask specific questions about additional surgery that has been done after the first surgery.
Number of patients with pelvic pain | +10 years after surgery
  Late complications due to surgery such as pelvic pain. We will send out questionnaires specifically asking about pelvic pain.
Number of participants with groin pain | +10 years after surgery
  Late complications due to surgery such as groin pain. We will send out questionnaires specifically asking about groin pain.
Number of participants with dyspareunia | +10 years after surgery
  Pain during sexual intercourse will be measured by the validated scale PISQ-12 (Pelvic Organ Prolapse/ Urinary Incontinence Sexual Questionnaire).
Number of participants that has had a reoperation | Up to 14 years after first surgery
  Reoperation due to complication after the first surgery. We will ask this in a questionnaire sent to all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Ek, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Obstetrics and Gynecology, Stockholm South General Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No